CLINICAL TRIAL: NCT01085227
Title: Clinical, Molecular and by Neuroimaging Characterization of Monogenic Forms of Parkinsonism Syndromes: Mutations of the LRRK2 Gene.
Brief Title: Clinical, Molecular and by Neuroimaging of LRRK2 Mutations
Acronym: LRRK2
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C06-16.1; 2007-A00169-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; LRRK2; asymptomatic carriers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients carrier of a LRRK2 mutation
- Asymptomatic relatives of LRRK2 patients

SUMMARY:
Besides Parkinson's disease (PD), it exists rare parkinsonian syndromes clinically close to PD and that correspond to Mendelian entities. Autosomal dominant forms are mainly associated with mutations of alpha synuclein and LRRK2/dardarin genes, whereas autosomal recessive forms are due to mutations in Parkin, Pink1 and DJ-1 genes. This entities are still unknown on the clinical, genetic and metabolic " au plan ".

Throughout a national network of 15 specialized centres in movement disorders, coordinated by the team of the neurogenetics reference centre at the Pitié-Salpêtrière Hospital (Alexis Brice), we propose to precise the relative frequency, the molecular bases and abnormalities in functional neuroimaging associated with the LRRK2 gene mutations, the most frequently implicated in the autosomal dominant forms. Due to the relative rarity of this parkinsonian syndrome, we will perform at the same time a retrospective study in cases and families already collected by the national network (300 isolated cases and 300 families) and a prospective study. The network will recruit 100 isolated cases and 40 familial cases yearly, with precise diagnosis tools. The genetic analysis will evaluate the relative frequency of the LRRK2 mutations and their spectrum in the French population. Phenotype-genotype correlations will be performed to better orientate the molecular diagnosis, in order to improve the genetic counselling and reduce costs of these analyses. In the case of LRRK2 mutations, a genetic investigation will be proposed to the families, with a specific care to at-risk cases. A detailed phenotypic evaluation of patients and at-risk cases will be proposed (neurological, neuropsychiatric and behavioural) at the CIC Pitié-Salpêtrière and also in imaging, for 15 patients and 40 of their relatives (20 carriers and 20 non-carriers of the LRRK2 mutation). The TEP study will evaluate the dopaminergic function (fluorodopa capture) and will measure the dopamine transporter (DAT). The structural MRI evaluation will search for possible associated structural morphologic abnormalities. The functional MRI evaluation will search for dysfunction of motor circuit during the movement realisation. These examinations will be performed at two years of interval for appreciate the evolution of the disease. This study will allow to better characterize the parkinsonian syndromes due to LRRK2 mutations and also to better characterize the presymptomatic phase, which is subject to controversies in idiopathic PD. The feasibility of this project is assured by the expertise of the collaborative centres and by the inclusion of a retrospective cohort, combined to a prospective cohort, which will allow to recruit sufficient patients and at-risk relatives for a rare genetic entity.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old
* Diagnosis of Parkinson's disease
* To be a first-degree relative to a LRRK2 patient
* Ability to understand the aim of the study
* Ability to sign the consent form

Exclusion Criteria:

* Non ability to understand the aim of the study
* Non ability to sign the consent form
* Inability to do a MRI
* Pregnant women or absence of an effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French population
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CEA - Service Hospitalier Frédéric Joliot, Orsay
  - Pitie-Salpetriere Hospital, Paris